CLINICAL TRIAL: NCT05987748
Title: The Clock Thickens: Morning or Evening Training for the Treatment of NAFLD? (TikTac Study)
Brief Title: The Clock Thickens: Morning or Evening Training for the Treatment of NAFLD?
Acronym: TikTac
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Maag Lever Darm Stichting (Other)
Responsible Party: Principal Investigator, Milena Schoenke, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83431.058.22
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Exercise; Circadian rhythms
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning exercise (Experimental): Individuals will exercise train at 8 AM three times per week for 12 weeks.
  Interventions: Behavioral: Exercise training
- Evening exercise (Experimental): Individuals will exercise train at 8 PM three times per week for 12 weeks.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Mixed exercise training containing strength and endurance elements carried out under supervision

SUMMARY:
The goal of this clinical trial is to investigate the different effect of morning and evening exercise training in individuals with non-alcoholic fatty liver disease (NAFLD). The main question it aims to answer is:

• Is morning or evening exercise better for the treatment of NAFLD?

Participants will follow a supervised exercise training program for three months with either morning or evening training and the effect on liver health will be assessed. Researchers will compare the morning to the evening exercise group to see if one training timepoint is more effective than the other in reducing the amount of fat in the liver and improving liver health.

DETAILED DESCRIPTION:
The aim of the study is to identify the effect of exercise timing on NAFLD. Additionally, we aim to increase the understanding of the exercise-related modulation of the metabolic and inflammatory processes causing NAFLD, including insulin resistance and dysbiosis of the gut microbiota. Forty obese patients with NAFLD will be enrolled by randomization to participate in an exercise training program over 12 weeks, either in the morning (n=20) or evening (n=20). Blood and stool samples will be collected before, during and after the intervention to monitor diagnostic markers such as liver enzymes (AST, ALT, GGT, etc.) and changes of the gut microbiota with exercise, respectively. Moreover, mixed meal tolerance tests will be performed before and after the intervention to monitor insulin sensitivity and hepatic fat content and cardiovascular parameters (e.g. arterial stiffness) will be monitored via MRI. Throughout the study, physical fitness will be assessed and monitored using steep ramp tests. Patients will be randomized for a supervised, standardized 50 min morning or evening training, with both progressive endurance and strength elements, in a frequency of 3 times a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years and ≤ 75
* Obese (BMI > 27 kg/m2)
* Males and postmenopausal females
* Caucasian
* Hepatic steatosis defined as increased hyperechogenicity of the liver on abdominal ultrasound, CAP score on Fibroscan > 280, and/or histological signs of steatosis
* Sedentary lifestyle (maximum of 20 minutes of moderate-to-vigorous physical activity per day on less than three days per week)
* Written informed consent

Exclusion Criteria:

* Exclusion criteria for MRI (claustrophobia, pacemaker, metal implants, etc.)
* Any other liver disease than NAFLD/NASH
* Present excessive alcohol use defined as > 2 units/day
* Recent use (< 3 months) of antibiotics
* Recent changes in dosages of regular medication (< 3 months)
* Recent (< 3 months) weight change (>5%)
* Recent (< 3 months) substantial diet changes
* Cardiovascular co-morbidity defined as heart failure, coronary insufficiency and hypertension in past history
* Comorbidity that contraindicates exercise training and exercise testing or that affects exercise response and exercise capacity
* Ongoing or recent use of glucocorticoids, oral/transdermal hormonal substitution, paclitaxel, theofyllin, amiodarone, myelosuppresive agents
* A psychiatric, addictive or any other disorder that compromises the subjects ability to understand the study content and to give written informed consent for participation in the study
* Working night or alternating shifts, known sleeping disorders such as narcolepsy or insomnia

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Liver fat content | 12 weeks
  Liver fat content (in %) will be measured by MRI LiverMultiScan

SECONDARY OUTCOMES:
Hepatic fibrosis | 12 weeks
  Hepatic stiffness (in kPa) will be measured as a proxy for liver fibrosis by Fibroscan (transient elastography)
Body mass index (BMI) | 12 weeks
  Body weight (in kg) and height (in m) will be combined to report BMI in kg/m^2
Fecal microbiota | 12 weeks
  Fecal microbiota composition assessed via microbial sequencing
Cardiorespiratory fitness | 12 weeks
  Peak workload (Wpeak) will be assessed with a the Steep Ramp Test (SRT) on a cycle ergometer
Waist circumference | 12 weeks
  Waist circumference (in cm) will be measured with a measuring tape
Blood pressure | 12 weeks
  Blood pressure (mmHg) will be measured using an arm cuff
Plasma levels of liver enzymes | 12 weeks
  Plasma levels of aspartate transaminase (ASAT), alanine aminotransferase (ALAT), gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP) (all in units/L) and bilirubin (in umol/L) will be quantified in the laboratory
Plasma insulin levels | 12 weeks
  Plasma insulin (in pmol/L) will be measured during a mixed meal test after 0, 10, 20, 30, 40, 60, 90, 120 and 180 minutes of the ingestion of a mixed meal
Plasma glucose levels | 12 weeks
  Plasma glucose (in mmol/L) will be measured during a mixed meal test after 0, 10, 20, 30, 40, 60, 90, 120 and 180 minutes of the ingestion of a mixed meal
Blood lipid levels | 12 weeks
  Blood triglyceride, LDL-cholesterol and HDL-cholesterol levels (all in mmol/L) will be quantified in the laboratory
Physical activity | 12 weeks
  Self-reported physical activity (minutes of moderate-intensity activity per week) will be assessed with the International Physical Activity Questionnaire (IPAQ)
Sleep | 12 weeks
  Sleeping habits (bedtime, time of falling asleep, time of waking up, sleep duration) will be assessed via the Munich Chronotype Questionnaire (MCTQs 5.0).
Food intake | 12 weeks
  Self-reported food intake (type of food, quantity, time of intake) will be assessed with 3-day food diaries

CONTACTS AND LOCATIONS:
Overall Officials: Milena Schönke, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Starting at publication
Access Criteria: IPD that underlie results in a publication will be made available upon reasonable request

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. Hepatology. 2018 Jan;67(1):123-133. doi: 10.1002/hep.29466. Epub 2017 Dec 1. PMID 28802062
- [Background] Stols-Goncalves D, Hovingh GK, Nieuwdorp M, Holleboom AG. NAFLD and Atherosclerosis: Two Sides of the Same Dysmetabolic Coin? Trends Endocrinol Metab. 2019 Dec;30(12):891-902. doi: 10.1016/j.tem.2019.08.008. Epub 2019 Oct 17. PMID 31630897
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Ruissen MM, Mak AL, Beuers U, Tushuizen ME, Holleboom AG. Non-alcoholic fatty liver disease: a multidisciplinary approach towards a cardiometabolic liver disease. Eur J Endocrinol. 2020 Sep;183(3):R57-R73. doi: 10.1530/EJE-20-0065. PMID 32508312
- [Background] Sato S, Basse AL, Schonke M, Chen S, Samad M, Altintas A, Laker RC, Dalbram E, Barres R, Baldi P, Treebak JT, Zierath JR, Sassone-Corsi P. Time of Exercise Specifies the Impact on Muscle Metabolic Pathways and Systemic Energy Homeostasis. Cell Metab. 2019 Jul 2;30(1):92-110.e4. doi: 10.1016/j.cmet.2019.03.013. Epub 2019 Apr 18. PMID 31006592
- [Background] Savikj M, Gabriel BM, Alm PS, Smith J, Caidahl K, Bjornholm M, Fritz T, Krook A, Zierath JR, Wallberg-Henriksson H. Afternoon exercise is more efficacious than morning exercise at improving blood glucose levels in individuals with type 2 diabetes: a randomised crossover trial. Diabetologia. 2019 Feb;62(2):233-237. doi: 10.1007/s00125-018-4767-z. Epub 2018 Nov 13. PMID 30426166
- [Background] Dalbram E, Basse AL, Zierath JR, Treebak JT. Voluntary wheel running in the late dark phase ameliorates diet-induced obesity in mice without altering insulin action. J Appl Physiol (1985). 2019 Apr 1;126(4):993-1005. doi: 10.1152/japplphysiol.00737.2018. Epub 2019 Feb 7. PMID 30730814
- [Background] Andersson A, Kelly M, Imajo K, Nakajima A, Fallowfield JA, Hirschfield G, Pavlides M, Sanyal AJ, Noureddin M, Banerjee R, Dennis A, Harrison S. Clinical Utility of Magnetic Resonance Imaging Biomarkers for Identifying Nonalcoholic Steatohepatitis Patients at High Risk of Progression: A Multicenter Pooled Data and Meta-Analysis. Clin Gastroenterol Hepatol. 2022 Nov;20(11):2451-2461.e3. doi: 10.1016/j.cgh.2021.09.041. Epub 2021 Oct 7. PMID 34626833
- [Background] Schaapman JJ, Tushuizen ME, Coenraad MJ, Lamb HJ. Multiparametric MRI in Patients With Nonalcoholic Fatty Liver Disease. J Magn Reson Imaging. 2021 Jun;53(6):1623-1631. doi: 10.1002/jmri.27292. Epub 2020 Aug 21. PMID 32822095
- [Background] Oeda S, Tanaka K, Oshima A, Matsumoto Y, Sueoka E, Takahashi H. Diagnostic Accuracy of FibroScan and Factors Affecting Measurements. Diagnostics (Basel). 2020 Nov 12;10(11):940. doi: 10.3390/diagnostics10110940. PMID 33198092
- [Background] Mikolasevic I, Orlic L, Franjic N, Hauser G, Stimac D, Milic S. Transient elastography (FibroScan((R))) with controlled attenuation parameter in the assessment of liver steatosis and fibrosis in patients with nonalcoholic fatty liver disease - Where do we stand? World J Gastroenterol. 2016 Aug 28;22(32):7236-51. doi: 10.3748/wjg.v22.i32.7236. PMID 27621571
- [Background] van Lingen E, Tushuizen ME, Steenhuis MEJ, van Deynen T, Martens J, Morales DD, van der Meulen-de Jong AE, Molendijk I, van der Marel S, Maljaars PWJ. Disease activity in inflammatory bowel disease patients is associated with increased liver fat content and liver fibrosis during follow-up. Int J Colorectal Dis. 2022 Feb;37(2):349-356. doi: 10.1007/s00384-021-04065-8. Epub 2021 Nov 17. PMID 34791524
- [Background] Beyer C, Hutton C, Andersson A, Imajo K, Nakajima A, Kiker D, Banerjee R, Dennis A. Comparison between magnetic resonance and ultrasound-derived indicators of hepatic steatosis in a pooled NAFLD cohort. PLoS One. 2021 Apr 1;16(4):e0249491. doi: 10.1371/journal.pone.0249491. eCollection 2021. PMID 33793651
- [Background] Dennis A, Mouchti S, Kelly M, Fallowfield JA, Hirschfield G, Pavlides M, Banerjee R. A composite biomarker using multiparametric magnetic resonance imaging and blood analytes accurately identifies patients with non-alcoholic steatohepatitis and significant fibrosis. Sci Rep. 2020 Sep 17;10(1):15308. doi: 10.1038/s41598-020-71995-8. PMID 32943694
- [Background] Amerikanou C, Kanoni S, Kaliora AC, Barone A, Bjelan M, D'Auria G, Gioxari A, Gosalbes MJ, Mouchti S, Stathopoulou MG, Soriano B, Stojanoski S, Banerjee R, Halabalaki M, Mikropoulou EV, Kannt A, Lamont J, Llorens C, Marascio F, Marascio M, Roig FJ, Smyrnioudis I, Varlamis I, Visvikis-Siest S, Vukic M, Milic N, Medic-Stojanoska M, Cesarini L, Campolo J, Gastaldelli A, Deloukas P, Trivella MG, Francino MP, Dedoussis GV; MAST4HEALTH consortium. Effect of Mastiha supplementation on NAFLD: The MAST4HEALTH Randomised, Controlled Trial. Mol Nutr Food Res. 2021 May;65(10):e2001178. doi: 10.1002/mnfr.202001178. Epub 2021 Apr 16. PMID 33629536
- [Background] Eilenberg M, Munda P, Stift J, Langer FB, Prager G, Trauner M, Staufer K. Accuracy of non-invasive liver stiffness measurement and steatosis quantification in patients with severe and morbid obesity. Hepatobiliary Surg Nutr. 2021 Oct;10(5):610-622. doi: 10.21037/hbsn-20-787. PMID 34760965
- [Background] Yang A, Nguyen M, Ju I, Brancatisano A, Ryan B, van der Poorten D. Utility of Fibroscan XL to assess the severity of non-alcoholic fatty liver disease in patients undergoing bariatric surgery. Sci Rep. 2021 Jul 7;11(1):14006. doi: 10.1038/s41598-021-93294-6. PMID 34234198
- [Background] Ciardullo S, Perseghin G. Statin use is associated with lower prevalence of advanced liver fibrosis in patients with type 2 diabetes. Metabolism. 2021 Aug;121:154752. doi: 10.1016/j.metabol.2021.154752. Epub 2021 Mar 11. PMID 33716004
- [Background] Kim D, Konyn P, Cholankeril G, Ahmed A. Physical Activity Is Associated With Nonalcoholic Fatty Liver Disease and Significant Fibrosis Measured by FibroScan. Clin Gastroenterol Hepatol. 2022 Jun;20(6):e1438-e1455. doi: 10.1016/j.cgh.2021.06.029. Epub 2021 Jun 29. PMID 34214678
- [Background] Albarazanji K, Nawrocki AR, Gao B, Wang X, Wang YJ, Xiao YF. Effects of mixed meal tolerance test on gastric emptying, glucose and lipid homeostasis in obese nonhuman primates. Sci Rep. 2021 Jun 4;11(1):11866. doi: 10.1038/s41598-021-91027-3. PMID 34088949
- [Background] Greenbaum CJ, Mandrup-Poulsen T, McGee PF, Battelino T, Haastert B, Ludvigsson J, Pozzilli P, Lachin JM, Kolb H; Type 1 Diabetes Trial Net Research Group; European C-Peptide Trial Study Group. Mixed-meal tolerance test versus glucagon stimulation test for the assessment of beta-cell function in therapeutic trials in type 1 diabetes. Diabetes Care. 2008 Oct;31(10):1966-71. doi: 10.2337/dc07-2451. Epub 2008 Jul 15. PMID 18628574
- [Background] Fujioka Y, Okura T, Sumi K, Matsumoto K, Shoji K, Nakamura R, Matsuzawa K, Izawa S, Kato M, Taniguchi S, Yamamoto K. Normal meal tolerance test is preferable to the glucagon stimulation test in patients with type 2 diabetes that are not in a hyperglycemic state: Comparison with the change of C-peptide immunoreactivity. J Diabetes Investig. 2018 Mar;9(2):274-278. doi: 10.1111/jdi.12692. Epub 2017 Jun 19. PMID 28494143
- [Background] Bacha F, Gungor N, Arslanian SA. Measures of beta-cell function during the oral glucose tolerance test, liquid mixed-meal test, and hyperglycemic clamp test. J Pediatr. 2008 May;152(5):618-21. doi: 10.1016/j.jpeds.2007.11.044. Epub 2008 Feb 4. PMID 18410762
- [Background] Hong Y, Dingemanse J, Sidharta P, Mager DE. Population pharmacodynamic modeling of hyperglycemic clamp and meal tolerance tests in patients with type 2 diabetes mellitus. AAPS J. 2013 Oct;15(4):1051-63. doi: 10.1208/s12248-013-9512-4. Epub 2013 Aug 1. PMID 23904152
- [Background] Carr RD, Larsen MO, Jelic K, Lindgren O, Vikman J, Holst JJ, Deacon CF, Ahren B. Secretion and dipeptidyl peptidase-4-mediated metabolism of incretin hormones after a mixed meal or glucose ingestion in obese compared to lean, nondiabetic men. J Clin Endocrinol Metab. 2010 Feb;95(2):872-8. doi: 10.1210/jc.2009-2054. Epub 2009 Dec 11. PMID 20008019
- [Background] Lages M, Barros R, Moreira P, Guarino MP. Metabolic Effects of an Oral Glucose Tolerance Test Compared to the Mixed Meal Tolerance Tests: A Narrative Review. Nutrients. 2022 May 12;14(10):2032. doi: 10.3390/nu14102032. PMID 35631171
- [Background] Wopereis S, Stroeve JHM, Stafleu A, Bakker GCM, Burggraaf J, van Erk MJ, Pellis L, Boessen R, Kardinaal AAF, van Ommen B. Multi-parameter comparison of a standardized mixed meal tolerance test in healthy and type 2 diabetic subjects: the PhenFlex challenge. Genes Nutr. 2017 Aug 29;12:21. doi: 10.1186/s12263-017-0570-6. eCollection 2017. PMID 28861127
- [Background] Meyer K, Samek L, Schwaibold M, Westbrook S, Hajric R, Beneke R, Lehmann M, Roskamm H. Interval training in patients with severe chronic heart failure: analysis and recommendations for exercise procedures. Med Sci Sports Exerc. 1997 Mar;29(3):306-12. doi: 10.1097/00005768-199703000-00004. PMID 9139168